CLINICAL TRIAL: NCT01259102
Title: A Parallel Open-Label Study to Examine Plasma Concentrations of Buprenorphine Following Reapplication of 10-mg Buprenorphine Transdermal System (BTDS) After Variable Application Site Rest Periods in Healthy Subjects
Brief Title: Examine Plasma Concentrations of Buprenorphine Following Reapplication of Buprenorphine Transdermal System (BTDS) After Variable Application Site Rest Periods
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: BUP1002
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2011-02-07 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Healthy subjects; Opioid; Transdermal
MeSH Terms: interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- No Rest (Experimental): BTDS 10 with no application site rest period prior to application of second BTDS
  Interventions: Drug: Buprenorphine transdermal patch
- 7-Day Rest (Experimental): BTDS 10 with 7-day rest period prior to application of second BTDS
  Interventions: Drug: Buprenorphine transdermal patch
- 14-Day Rest (Experimental): BTDS 10 with 14-day rest period prior to application of second BTDS
  Interventions: Drug: Buprenorphine transdermal patch
- 21-Day Rest (Experimental): BTDS 10 with 21-day rest period prior to application of second BTDS
  Interventions: Drug: Buprenorphine transdermal patch
- 28-Day Rest (Experimental): BTDS 10 with 28-day rest period prior to application of second BTDS
  Interventions: Drug: Buprenorphine transdermal patch

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine 10 mcg/hour patch applied transdermally for 7-day wear.
  Other Names: Butrans™

SUMMARY:
The purpose of this study is to determine the pharmacokinetics of BTDS following same-site patch reapplication after rest intervals.

DETAILED DESCRIPTION:
The purpose of this study is to determine the minimum application site rest period that ensures that reapplication of BTDS 10 to the same site in the deltoid region does not result in increased absorption of drug in normal healthy subjects.

ELIGIBILITY:
Inclusion Criteria Include:

* Males and females 18 to 45 years of age, inclusive.
* Weight of 60 to 100 kilograms (kg) [132-220 pounds (lb)] and within 15% of optimum for height and body frame.
* In good health, evidenced by a lack of significantly abnormal findings on medical history, physical examination, clinical laboratory tests, vital signs, and electrocardiogram (ECG).
* Willing to discontinue and abstain from any medications, including vitamins or mineral supplements, throughout the study.
* Willing to follow dietary restrictions, including abstention from caffeine and xanthine-containing beverages for the duration of the study.
* Did not smoke or chew tobacco for at least 45 days prior to administration of study drugs, and agree not to use tobacco products during the study

Exclusion Criteria Include:

* A history of hypersensitivity to opioid or psychotropic drugs.
* A history of recurrent seizures or syncope.
* Any medical or surgical conditions which might interfere with transdermal absorption, distribution, metabolism, or excretion of drugs.
* Any other significant active medical illness such as: history or presence of liver disease or liver injury that is indicated by an abnormal liver function profile such as aspartate transaminase (AST), alanine transaminase (ALT), or serum bilirubin; history or presence of impaired renal function that is indicated by abnormal creatinine or blood urea nitrogen (BUN) values or abnormal urinary constituents (eg, albuminuria); history of neutropenia (absolute neutrophil count [ANC] <1000/mm3 or thrombocytopenia (platelet <150,000/mm3).
* Positive results of urine drug screen or urine cotinine (consistent with active smoking).
* A history of substance or alcohol abuse within the past 5 years.
* Females who are nursing.
* Females who are pregnant as confirmed by a positive serum human chorionic gonadotropin (bHCG) test.

Other protocol-specific exclusion/inclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2000-11; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Department of Pharmacology, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19-Nov-2000 (first patient, first visit) to 18-Mar-2001 (last patient, last visit) at 1 center in the US, Columbus, OH.
Pre-assignment Details: Subjects were assigned into 1 of 5 treatment groups with different recovery periods, ranging from 0 to 4 weeks. For the 5 treatment groups, the rest period was 0, 7, 14, 21, or 28 days, respectively, between the removal of the first buprenorphine transdermal system (BTDS) and placement of the second BTDS in exactly the same location.
Groups:
- No Rest: Each subject applied BTDS (10 mcg/h) on 2 occasions and wore it for 7 days (168 hours). Subjects were assigned to 1 of 5 treatment groups with different application site rest periods from 0 to 4 weeks. For this group, the rest period was 0 days between the removal of BTDS and placement of the second BTDS in the same location.
- 7-Day Rest: Each subject applied BTDS (10 mcg/h) on 2 occasions and wore it for 7 days (168 hours). Subjects were assigned to 1 of 5 treatment groups with different application site rest periods from 0 to 4 weeks. For this group, the rest period was 7 days between the removal of BTDS and placement of the second BTDS in the same location.
- 14-Day Rest: Each subject applied BTDS (10 mcg/h) on 2 occasions and wore it for 7 days (168 hours). Subjects were assigned to 1 of 5 treatment groups with different application site rest periods from 0 to 4 weeks. For this group, the rest period was 14 days between the removal of BTDS and placement of the second BTDS in the same location.
- 21-Day Rest: Each subject applied BTDS (10 mcg/h) on 2 occasions and wore it for 7 days (168 hours). Subjects were assigned to 1 of 5 treatment groups with different application site rest periods from 0 to 4 weeks. For this group, the rest period was 21 days between the removal of BTDS and placement of the second BTDS in the same location.
- 28-Day Rest: Each subject applied BTDS (10 mcg/h) on 2 occasions and wore it for 7 days (168 hours). Subjects were assigned to 1 of 5 treatment groups with different application site rest periods from 0 to 4 weeks. For this group, the rest period was 28 days between the removal of BTDS and placement of the second BTDS in the same location.
Period: Overall Study
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Started | 13 | 14 | 15 | 14 | 14
Completed | 12 | 14 | 13 | 12 | 13
Not Completed | 1 | 0 | 2 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest | Total
Number analyzed (Participants) | 13 | 14 | 15 | 14 | 14 | 70
Age Continuous [Mean (Standard Deviation); unit: years] | 28.8 (1.9) | 26.2 (1.6) | 23.3 (1.1) | 26.4 (1.9) | 25.1 (2.3) | 25.9 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 1 | 0 | 4
  Male | 11 | 14 | 14 | 13 | 14 | 66
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 3 | 0 | 1 | 0 | 3 | 7
  Black or African American | 4 | 3 | 1 | 1 | 2 | 11
  White | 6 | 9 | 13 | 12 | 9 | 49
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Period 1: AUC0-3d
Description: Period 1 was the first application of BTDS 10: To determine the minimum application site rest periods that ensured that the reapplication of BTDS to the same site in the deltoid region did not result in increased absorption of the drug as measured by AUC0-3d [The area under the plasma concentration-time course profile from time = 0 (dosing) through day 3 (to 72 hours)].
Time Frame: 0 to 3 days (72 hours)
Population: Pharmacokinetic Population: All subjects who satisfied the inclusion/exclusion criteria, received both applications of BTDS, and submitted to postbaseline phlebotomy through at least the 72-hour time point of both applications.
Measure: Mean (Standard Error); unit: pg/mL*h
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
pg/mL*h | 8680 (920) | 7651 (1514) | 6465 (1091) | 12258 (836) | 8890 (1054)

2. Primary Outcome: Period 2: AUC0-3d.
Description: Period 2 was the second application of BTDS 10: To determine the minimum application site rest periods that ensured that the reapplication of BTDS to the same site in the deltoid region did not result in increased absorption of the drug as measured by AUC0-3d.
  AUC0-3d - The area under the plasma concentration-time course profile from time = 0 (dosing) through day 3 (to 72 hours).
Time Frame: 0 to 3 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL*h
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
pg/mL*h | 12316 (1062) | 14733 (2255) | 13571 (1671) | 12931 (908) | 9056 (888)

3. Primary Outcome: Period 1: Cmax0-3d
Description: Period 1 was the first application of BTDS 10: To determine the minimum application site rest periods that ensured that the reapplication of BTDS to the same site in the deltoid region did not result in increased absorption of the drug as measured by Cmax0-3d.
  Cmax0-3d - The maximum observed concentration taken directly from the plasma concentration-time course profile from time = 0 (dosing) through day 3 (to 72 hours). This was considered an index of maximum (peak) exposure to the study drug.
Time Frame: 0 to 3 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
pg/mL | 183 (17) | 193 (50) | 151 (24) | 241 (15) | 185 (16)

4. Primary Outcome: Period 2: Cmax0-3d
Description: Period 2 was the second application of BTDS 10: To determine the minimum application site rest periods that ensured that the reapplication of BTDS to the same site in the deltoid region did not result in increased absorption of the drug as measured by Cmax0-3d.
  Cmax0-3d (pg/mL) - The maximum observed concentration taken directly from the plasma concentration-time course profile from time = 0 (dosing) through day 3 (to 72 hours). This was considered an index of maximum (peak) exposure to the study drug.
Time Frame: 0 to 3 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
pg/mL | 216 (17) | 300 (52) | 262 (31) | 278 (41) | 182 (14)

5. Secondary Outcome: Period 1: AUC0-7d.
Description: Period 1 was the first application of BTDS 10: The time for absorption to return to normal measured by AUC0-7d.
  AUC0-7d - The area under the plasma concentration-time course profile from time = 0 (dosing) to BTDS removal.
Time Frame: 0 to 7 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL*h
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
pg/mL*h | 21946 (1686) | 20541 (2645) | 14707 (1851) | 27040 (1298) | 22086 (1591)

6. Secondary Outcome: Period 2: AUC0-7d
Description: Period 2 was the second application of BTDS 10: The time for absorption to return to normal measured by AUC0-7d.
  AUC0-7d - The area under the plasma concentration-time course profile from time = 0 (dosing) to BTDS removal.
Time Frame: 0 to 7 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL*h
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
pg/mL*h | 25126 (2285) | 27543 (3093) | 26174 (2414) | 27123 (1475) | 21790 (1365)

7. Secondary Outcome: Period 1: Cmax0-7
Description: Period 1 was the first application of BTDS 10: The time for absorption to return to normal measured by Cmax0-7.
  Cmax0-7d - The maximum observed concentration taken directly from the plasma concentration-time course profile.
Time Frame: 0 to 7 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
pg/mL | 188 (16) | 206 (48) | 160 (22) | 245 (14) | 192 (15)

8. Secondary Outcome: Period 2: Cmax0-7d
Description: Period 2 was the second application of BTDS 10: The time for absorption to return to normal measured by Cmax0-7d.
  Cmax0-7d - The maximum observed concentration taken directly from the plasma concentration-time course profile.
Time Frame: 0 to 7 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
pg/mL | 216 (17) | 300 (52) | 262 (31) | 278 (41) | 202 (18)

9. Secondary Outcome: Period 1: Tmax0-7d.
Description: Period 1 was the first application of BTDS 10: The time for absorption to return to normal measured by Tmax0-7d.
  Tmax0-7d - The time from dosing to the maximum observed concentration was taken directly from the plasma concentration-time course profile. If the maximum plasma concentration was observed at 2 or more consecutive time points, the earliest time point was used for Tmax.
Time Frame: 0 to 7days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: hour
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
hour | 74 (7) | 86 (6) | 78 (15) | 55 (6) | 76 (11)

10. Secondary Outcome: Period 2: Tmax0-7d.
Description: Period 2 was the second application of BTDS 10: The time for absorption to return to normal measured by Tmax0-7d.
  Tmax0-7d - The time from dosing to the maximum observed concentration was taken directly from the plasma concentration-time course profile. If the maximum plasma concentration was observed at 2 or more consecutive time points, the earliest time point was used for Tmax.
Time Frame: 0 to 7 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: hour
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Number analyzed (Participants) | 12 | 11 | 13 | 12 | 12
hour | 42 (3) | 38 (6) | 36 (5) | 46 (4) | 63 (10)

ADVERSE EVENTS:
Time Frame: All adverse events, whether spontaneously reported or elicited on direct questioning, that occurred after administration of the first dose of study drug and on or before the final visit were reported on the adverse event form.
Description: AEs were learned of by spontaneous reports and subject interview.
Arm/Group | No Rest | 7-Day Rest | 14-Day Rest | 21-Day Rest | 28-Day Rest
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/14 | 0/15 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 11/13 | 14/14 | 13/15 | 10/14 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Rest (N=13) | 7-Day Rest (N=14) | 14-Day Rest (N=15) | 21-Day Rest (N=14) | 28-Day Rest (N=14)
Neutropenia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | No Rest (N=13) | 7-Day Rest (N=14) | 14-Day Rest (N=15) | 21-Day Rest (N=14) | 28-Day Rest (N=14)
Phlebitis (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Anorexia (Gastrointestinal disorders) | 4 | 5 | 2 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 7 | 3 | 7 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2
Asthenia (General disorders) | 7 | 2 | 4 | 0 | 2
Headache (General disorders) | 6 | 8 | 10 | 1 | 6
Thirst (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 0 | 1
Nervousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Thinking abnormally (Psychiatric disorders) | 1 | 1 | 0 | 2 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3
Prutitus at site (Skin and subcutaneous tissue disorders) | 5 | 0 | 3 | 0 | 2
Polyuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Accidental injury (General disorders) | 0 | 1 | 0 | 0 | 0
Back pain (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain substernal (General disorders) | 1 | 0 | 0 | 0 | 0
Infection (General disorders) | 0 | 0 | 0 | 1 | 0
Infection bacterial (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 1
Reaction unevaluable (General disorders) | 1 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Palpitation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Vasodilatation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Bilirubinemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Agitation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 5 | 5 | 5 | 5 | 5
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cough increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Erythema at site (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Other site reactions (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Amblyopia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 1 | 0 | 0
Abnormal ejaculation (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days